CLINICAL TRIAL: NCT01983306
Title: A Randomized, 4-Week, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Assess the Safety and Efficacy of SP-333 for the Treatment of Opioid-induced Constipation (OIC) in Patients With Non-malignant Chronic Pain Receiving Opioid Therapy
Brief Title: Dose-ranging Study to Assess Safety and Efficacy of SP-333 for the Treatment of Opioid-induced Constipation (OIC)
Acronym: OIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP333201-01
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Constipation
Keywords: Constipation; Opioid; GC C Agonist; Pain
MeSH Terms: conditions — Constipation; Pain | interventions — dolcanatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SP-333 1 mg (Experimental): 1 mg SP-333 orally once daily for 4-week Treatment Period
  Interventions: Drug: SP-333 1 mg
- SP-333 3 mg (Experimental): 3 mg SP-333 orally once daily for 4-week Treatment Period
  Interventions: Drug: SP-333 3 mg
- SP-333 6 mg (Experimental): 6 mg SP-333 orally once daily for 4-week Treatment Period
  Interventions: Drug: SP-333 6 mg
- Placebo (Placebo Comparator): Placebo orally once daily for 4-week Treatment Period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-333 1 mg — Tablet
  Arms: SP-333 1 mg
Drug: SP-333 3 mg — Tablet
  Arms: SP-333 3 mg
Drug: SP-333 6 mg — Tablet
  Arms: SP-333 6 mg
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a range of oral SP-333 doses for the treatment of opioid-induced constipation (OIC) in adults with non-cancer pain taking opioids.

ELIGIBILITY:
Inclusion Criteria:

* Must be receiving chronic, stable opioid therapy to treat non-malignant pain for at least 3 months prior to screening
* Must have active OIC at screening
* Active OIC must be confirmed during baseline screening bowel habit and symptom diary
* Must be on stable diet

Exclusion Criteria:

* Has history of chronic therapy for chronic constipation prior to start of opioid therapy, or any potential non-opioid cause of bowel dysfunction that may be a major contributor to the constipation (i.e., mechanical obstruction or pseudo-obstruction)
* Use of medications that might affect bowel movement frequency or constipation-related symptoms (e.g., prokinetics, anti-diarrheal agents, laxatives other than study-defined rescue laxative)
* Has history of or current cancer (other than basal cell or squamous cell carcinoma of the skin) unless the malignancy has been in complete remission without maintenance chemotherapy for at least 5 years
* Unstable thyroid disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of spontaneous bowel movements during Week 4 of the 4-week treatment period | 4 Weeks
  Compare SP-333 (1, 3 & 6 mg) with placebo in the treatment of OIC as measured by the change from baseline in the number of spontaneous bowel movements during Week 4 of the 4-week treatment period

SECONDARY OUTCOMES:
To assess safety and tolerability of SP-333 in the treatment of non-malignant OIC | 4 weeks
  Compare the safety and tolerability of SP-333 (1, 3 & 6 mg) with placebo as measured by rates of adverse events, clinical laboratory abnormalities and significant changes in vital signs and ECGs.

OTHER OUTCOMES:
To evaluate stool consistency over the 4-week Treatment Period | 4 weeks
  Compare SP-333 (1, 3 & 6 mg) with placebo in rates of change from baseline in stool consistency over the 4 weeks of treatment.
To evaluate constipation-related symptoms over the 4-week Treatment Period | 4 weeks
  Compare SP-333 (1, 3 & 6 mg) with placebo in rates of change from baseline in constipation-related symptoms over the 4 weeks of treatment.
To evaluate bowel movement frequency responder rates [Complete Spontaneous Bowel Movements (CSBMs) and Spontaneous Bowel Movements (SBMs)] over the 4-week Treatment Period. | 4 weeks
  Compare SP-333 (1, 3 & 6 mg) with placebo in rates of change from baseline for bowel movement frequency responder rates [Complete Spontaneous Bowel Movements (CSBMs) and Spontaneous Bowel Movements (SBMs)] over the 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Tenenbaum, Study Director — Synergy Pharmaceuticals Inc.
Locations (38):
- United States (38):
  - Synergy Research Site, Huntsville, Alabama
  - Synergy Research Site, Mobile, Alabama
  - Synergy Research Site, Phoenix, Arizona
  - Synergy Research Site, Artesia, California
  - Synergy Research Site, Laguna Hills, California
  - Synergy Research Site, Oceanside, California
  - Synergy Research Site, Sacramento, California
  - Synergy Research Site, San Diego, California
  - Synergy Research Site, San Francisco, California
  - Synergy Research Site, Hialeah, Florida
  - Synergy Research Site, Miami, Florida
  - Synergy Research Site, Miami Beach, Florida
  - Synergy Research Site, Plant City, Florida
  - Synergy Research Site, Plantation, Florida
  - Synergy Research Site, Port Orange, Florida
  - Synergy Research Site, Sarasota, Florida
  - Synergy Research Site, West Palm Beach, Florida
  - Synergy Research Site, Winter Haven, Florida
  - Synergy Research Site, Atlanta, Georgia
  - Synergy Research Site, Bloomington, Illinois
  - Synergy Research Site, Traverse City, Michigan
  - Synergy Research Site, St Louis, Missouri
  - Synergy Research Site, Las Vegas, Nevada
  - Synergy Research Site, Great Neck, New York
  - Synergy Research Site, New York, New York
  - Synergy Research Site, Concord, North Carolina
  - Synergy Research Site, Greensboro, North Carolina
  - Synergy Research Site, Salisbury, North Carolina
  - Synergy Research Site, Winston-Salem, North Carolina
  - Synergy Research Site, Dayton, Ohio
  - Synergy Research Site, Oklahoma City, Oklahoma
  - Synergy Research Site, Medford, Oregon
  - Synergy Research Site, Orangeburg, South Carolina
  - Synergy Research Site, Chattanooga, Tennessee
  - Synergy Research Site, Arlington, Texas
  - Synergy Research Site, Dallas, Texas
  - Synergy Research Site, Houston, Texas
  - Synergy Research Site, San Antonio, Texas